CLINICAL TRIAL: NCT05384314
Title: A Retrospective Study to Evaluate the Predictability of Abnormal Arterial Blood Gas Measurements Through Novel Observations of Continuous Trends in Electronically Measured Respiratory Rate in a Mixed Cohort of Respiratory Compromised Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor of Respiratory Medicine, Beaumont Hospital
Other Study IDs: RespiraSense ABG investigation
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Failure; COPD; Pneumonia; Community-acquired Pneumonia; COVID-19; Pulmonary Disease
Keywords: Respiratory Rate; Arterial Blood Gas
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Pneumonia; Community-Acquired Pneumonia; COVID-19; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Patients admitted with COPD as the primary admission.
  Interventions: Device: RespiraSense
- Respiratory Compromised General: Patients admitted with Pneumonia, COPD, COVID, to be included
  Interventions: Device: RespiraSense

INTERVENTIONS:
Device: RespiraSense — The use of continuous electronic monitoring of respiratory rate

SUMMARY:
A retrospective study to evaluate the predictability of abnormal arterial blood gas measurements through novel observations of continuous trends in electronically measured respiratory in a mixed cohort of respiratory compromised patients.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory condition is the primary admission diagnosis

Exclusion Criteria:

* Pregnant patients in their 2nd or 3rd trimester

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted respiratory compromised patients in a hospital setting
Sampling Method: Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-10-12 (Estimated); Study Completion 2022-12-12 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value/Precision (PPV) | 12 months
  Positive Predictive Value/Precision (PPV) of an elevated RespiraSense monitoring Respiratory Rate (RR) for an abnormal ABG - for a single disease state (COPD)

SECONDARY OUTCOMES:
PPV of an elevated RR for an abnormal ABG - for a mix of disease states | 12 months
  PPV of an elevated RR for an abnormal ABG - for a mix of disease states, all of which fall under Respiratory Failure

OTHER OUTCOMES:
PPV of elevated RR | 6 months
  PPV of elevated RR (for each of i. and ii. above) for requirement of a meaningful intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available.